CLINICAL TRIAL: NCT00742066
Title: Insulin-induced Microvascular Activity in Patients With Essential Hypertension: a Possible Role for Angiotensin II AT1-receptor Blockers.
Brief Title: Role of AT1-receptor Blockers in Insulin-induced Vasodilation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Prof. CDA Stehouwer, University Hospital Maastricht
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MEC 07-2-115
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Hypertension; Insulin Resistance; Microcirculation
Keywords: Hypertension; Insulin resistance; Microcirculation; Angiotensin II receptor blocker
MeSH Terms: conditions — Hypertension; Insulin Resistance | interventions — Irbesartan; Felodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- I (Experimental): Irbesartan
  Interventions: Drug: Irbesartan
- II (Active Comparator): Felodipine
  Interventions: Drug: Felodipine
- III (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Irbesartan — Single dose 600mg orally
  Other Names: Aprovel C09CA04
  Arms: I
Drug: Felodipine — single dose 10mg Felodipine ER
  Other Names: Plendil C08CA02
  Arms: II
Drug: Placebo — Single dose tablet orally
  Arms: III

SUMMARY:
In this study we hypothesize that blocking the angiotensin II AT1-receptor improves the insulin-induced microvascular dilatation. Objectives: 1. Does blockade of the angiotensin II AT1-receptor improve the insulin-induced microvascular effects in hypertensive patients. 2. Does blockade of the angiotensin II AT1-receptor impair the insulin-induced microvascular effects in normotensive control subjects?

ELIGIBILITY:
Inclusion Criteria:

hypertensive subjects:

1. 18-60 years
2. Caucasian
3. untreated hypertension >140/90mmHg.

normotensive subjects:

1. 18-60 years
2. Caucasian
3. Blood pressure <140/90 mmHg.

Exclusion Criteria:

1. Obesity (BMI>27kg/m2)
2. Cardiovascular disease (stroke, coronary artery disease, peripheral vascular disease, heart failure)
3. Impaired glucose tolerance or diabetes mellitus according to the criteria of the ADA
4. Smoking
5. Alcohol use >4U/day
6. Use of medication (antihypertensive drugs, lipid lowering drugs, corticosteroids, NNSAIDs)
7. Pregnancy
8. Wearing contact lenses

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
functional recruitment of capillaries in the skin | July 2009

SECONDARY OUTCOMES:
perfused capillary density in the nailfold | July 2009
Endothelium- (in)dependent vasodilatation of finger skin microcirculation | July 2009
Density of arterioles, capillaries and venules in the bulbar conjunctiva. | July 2009
Diameter of arterioles and venules in the bulbar conjunctiva | July 2009

CONTACTS AND LOCATIONS:
Overall Officials: CDA Stehouwer, Prof., Study Chair — Univeristy Hospital Maastricht
Locations (1):
- University Hospital Maastricht, Maastricht, P.O. Box 5800, Netherlands